CLINICAL TRIAL: NCT07341165
Title: Regulation of Satellite Cells and Myogenesis in Response to Eccentric Resistance Exercise in Hypoxic Conditions in Healthy Young Men
Brief Title: Regulation of Satellite Cells and Myogenesis in Response to Eccentric Resistance Exercise in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SCHYPECC
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Exercise; Hypoxia; Satellite Cells; Myogenesis
MeSH Terms: conditions — Motor Activity; Hypoxia | interventions — Blood Specimen Collection; Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance exercise in normoxia (Active Comparator): Group that performed the resistance exercise in normoxia (FiO2=0.21)
  Interventions: Device: Resistance exercise on an isokinetic dynamometer; Procedure: Vastus lateralis biopsy; Procedure: Blood samples; Device: Normoxia
- Resistance exercise in hypoxia (Experimental): Group that performed the resistance exercise in hypoxia (FiO2=0.14)
  Interventions: Device: Resistance exercise on an isokinetic dynamometer; Procedure: Vastus lateralis biopsy; Procedure: Blood samples; Device: Hypoxia
- Resistance exercise with blood flow restriction (Experimental): Group that performed the resistance exercise with blood flow restriction (60%AOP)
  Interventions: Device: Resistance exercise on an isokinetic dynamometer; Procedure: Vastus lateralis biopsy; Procedure: Blood samples; Device: Blood flow restriction

INTERVENTIONS:
Device: Resistance exercise on an isokinetic dynamometer — Leg flexion/extension: 5 series of 15 repetitions at 60°/sec for the knee extension and 30°/sec for the knee flexion
Procedure: Vastus lateralis biopsy — Biopsy taken in the vastus lateralis
Procedure: Blood samples — Blood samples taken from the antecubital vein
Device: Normoxia — Environmental condition for exercise: in a pressurized chamber with a inspired oxygen fraction of 0.21 (sea level)
  Arms: Resistance exercise in normoxia
Device: Hypoxia — Environmental hypoxia: in a chamber where oxygen is extracted and replaced by nitrogen to reach an inspired oxygen fraction of 0.135 (equivalent to 2500m altitude)
  Arms: Resistance exercise in hypoxia
Device: Blood flow restriction — Tourniquet placed around the proximal extremity of the lower limb and inflated at 60% of arterial occlusion pressure to induce local hypoxia
  Arms: Resistance exercise with blood flow restriction

SUMMARY:
Satellite cells (SC) are muscle stem cells that once activated, proliferate, and differentiate into myocytes that finally fuse with an existing myofiber to regenerate or increase its mass. This process is called 'myogenesis'. Satellite cell activation can be modulated by exercise and by hypoxia. Hypoxia is a state of lower availability of oxygen that can be reached either by going at high altitude (hypobaric hypoxia) or by lowering the percentage of oxygen in hypoxic rooms at sea level. In opposition to the previously described systemic hypoxia, local hypoxia can be reached placing a cuff around a limb, which will induce a partial vascular occlusion. The latter is termed as blood flow restriction (BFR). In addition, in response to physical exercise, a local intramuscular hypoxia can be found back in the skeletal muscle. Myogenesis has been shown to be modulated by hypoxia in different ways, depending on the level of hypoxia: in conditions of mild hypoxia, satellite cell proliferation appears to be favorized, whereas SC differentiation is decreased in those conditions. In conditions of severe hypoxia, SC quiescence is promoted. SC activation increases in response to resistance training, with and without BFR. Some recent data also suggest that resistance exercise in hypoxic rooms may modulate SC activation, but this area is less well understood. Eccentric exercise may enhance SC activation in comparison to concentric contraction. Up to now, no study has analyzed SC activation and myogenesis in response to an eccentric exercise in hypoxia. Whereas macroscopic differences such as higher muscle force gains or hypertrophy, have been observed between normoxic and hypoxic resistance training, but could not be explained by the classical protein balance and growth factors, there is a need for a better understanding of the muscle response in hypoxia and several studies suggest a role of satellite cells and myogenesis in that difference. The purpose of this study is to elucidate whether or not satellite cells are regulated in a different way in response to an eccentric exercise in hypoxia comparing to normoxia. In addition, differences in SC activation between environmental normobaric hypoxia and BFR, two methods used to reach hypoxia at sea level, are not well understood yet. Finally, most of the studies evaluating myogenic response following a resistance exercise have only taken samples at two time-points, before and 24h after exercise in most of the cases. As the different steps of the myogenic process evolves over the days and may be enhanced or inhibited by hypoxic conditions, multiple time-points would be interesting to observe the evolution of the myogenic process. In that purpose, blood and skeletal muscle samples will be taken at different time-points to evaluate the progress of myogenesis following an acute eccentric exercise. Myogenic regulatory factors will be analyzed by RT-qPCR (mRNA), Western-Blot (protein) and immunofluorescence (localization). In addition, factors able to regulate myogenesis such as muscle damage, inflammation, growth factors, early-regulated genes, MAPK… will also be analyzed in order to understand if they play a role in response to hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man
* Aged between 20 and 49 years
* Physically active
* Not involved in resistance training,
* No exposed to high altitude (>1500m) 1 month before experiment

Exclusion Criteria:

* Intake of AINS,
* Illness with altered inflammatory status,
* Condition that prohibits resistance exercise (muscle injury) or the sampling of tissue biopsies (aspirin, anticoagulants, allergy to lidocaine)

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Analysis of markers of satellite cells and myogenesis | Throughout the entire study, approximately during 30 months

SECONDARY OUTCOMES:
Comparison of the differences between exercise in environmental and local hypoxia | Throughout the entire study, approximately during 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculté des Sciences de la Motricité, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No